CLINICAL TRIAL: NCT06606041
Title: Comparison of the Efficacy of Dry Needling, Ischemic Compression, and Cross Taping on Masseter Myofascial Pain: A Randomized Clinical Trial
Brief Title: Comparison of the Efficacy of Dry Needling, Ischemic Compression, and Cross Taping on Masseter Myofascial Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Bruno Macedo de Sousa, Professor, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMUC-MD-PAIN
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Temporomandibular Joint Disorders; Myofascial Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Dry Needling; Acupressure

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized parallel clinical trial comparing Dry Needling, Ischemic Compression, and Cross Tapes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator)
  Interventions: Procedure: Dry Needling
- Group 2 (Active Comparator)
  Interventions: Procedure: Ischemic Compression
- Group 3 (Active Comparator)
  Interventions: Procedure: Cross Tapes

INTERVENTIONS:
Procedure: Dry Needling — This. minimally invasive technique is based on the insertion of a sterile, low-caliber, monofilament needle, without the injection or extraction of any additional substances, into hyperirritable muscle nodules. There are two categories within this technique, based on the depth at which the needle is inserted: superficial needling (or the Baldry technique), in which the needle is inserted up to the subcutaneous cellular tissue overlying the myofascial trigger point (up to 10 mm); and deep needling, where the needle is inserted into the muscle with the intention of reaching the myofascial trigger point. Reaching the trigger point was the investigators goal. Regardless of the technique selected, the aim is to generate controlled micro spasms in the affected muscle area, alternating with periods of muscle relaxation.
  Arms: Group 1
Procedure: Ischemic Compression — Ischemic compression is a conservative, manual technique used on myofascial trigger points, in which pressure should be exerted between 30 and 90 seconds on these same areas. It is suggested that it leads to the normalization of the biomechanical properties of muscle fibers, restoring the muscle's functional condition and probably reducing the risk of injury. Thus, the therapeutic effects include the stimulation of mechanoreceptors, with pain attenuation mainly due to the depletion of specific neurotransmitters and temporary obstruction of local blood flow (local ischemia), followed by a rapid influx of oxygenated blood to the area under pressure relief,(37) which will cause an increase in muscle metabolism.
  Arms: Group 2
Procedure: Cross Tapes — Cross tapes, as the name implies, based on an equidistant intersection of three or four polyester tapes with a non-elastic adhesive acrylic coating, with the 3 lines oriented in a latero-medial direction. It is recommended that it be applied to the muscle area where the myofascial trigger point has been detected, at a 45º angle to the muscle fibers. Its application may have several purposes, such as muscle support, improving the stability of the fibers; pain relief, especially in areas where muscle tension and/or inflammation are present; aiding lymphatic drainage; promoting blood circulation. Before it is applied, the skin should be clean (disinfecting the area with alcohol) and dry, without any lotion or other ointments and the maximum period of use should not exceed 24 hours due to the risk of changes in position, either due to sweating or direct intervention by the patient himself.
  Arms: Group 3

SUMMARY:
The goal of this clinical trial is to learn whether Dry Needling, Ischemic Compression, and Cross Tapes work to treat myofascial pain in masseter muscles in adults. It will also learn about the safety of this treatment. The main questions it aims to answer are:

* Do Dry Needling, Ischemic Compression, and Cross Tapes relieve masseter muscle pain?
* Which of these treatments provides the best relief from masseter muscle pain? Researchers will compare these three treatments to see which is best for treating masseter muscle pain.

Participants will:

Treated with Dry Needling or Ischemic Compression or Cross Tapes only once Visit the clinic one week, three months, and six months after treatment.

DETAILED DESCRIPTION:
The taut band represents the most commonly observed muscular disorder, where myofascial trigger points may arise, causing referred pain in another location. Therapeutic strategies applied for its treatment include dry needling, ischemic compression, and cross-taping.

Objectives: To compare the effectiveness of these treatment methods in reducing or alleviating the intensity of pain in the masseter.

In this multicenter randomized clinical trial, the study sample underwent a clinical examination according to the Diagnostic Criteria for Temporomandibular Disorders to diagnose the presence of orofacial myofascial pain with taut bands in the masseter. Participants were randomly allocated to three groups based on the treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myofascial pain diagnosed according Diagnostic Criteria for Temporomandibular Disorders (DC-TMD).

Exclusion Criteria:

* Pregnant women
* Other TMD-spectrum pathologies
* Anticoagulated and antiaggregated individuals
* Diabetes
* Blood disorders
* Fibromyalgia
* Autoimmune diseases in acute stages
* Neurological diseases
* Malignant tumor pathologies
* Patients with aichthyophobia
* Concomitant medication (opioids, antidepressants, myorelaxants)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At baseline, immediately after the intervention, 1 week, and 1 month after treatment
  Pain intensity will be assessed using the Numerical Pain Rating Scale, where 0 represents the absence of pain, and 10 describes the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Maria João Rodrigues, PhD, Study Chair — Faculty of Medicine, Institute of Occlusion and Orofacial Pain, University of Coimbra
Locations (2):
- Faculty of Medicine, Institute of Occlusion and Orofacial Pain, University of Coimbra, Coimbra, Portugal
- Faculty of Medicine of the University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No